CLINICAL TRIAL: NCT01713374
Title: Studies on the Physiological Meaning of Flow-mediated Constriction, Flow-mediated Dilatation and Vasomotion/Flowmotion: Circadian Variability and Role of the Sympathetic Nervous System.
Brief Title: Physiological Assessment of the Endothelium - Circadian Rhythm and Role of the Sympathetic Nervous System
Acronym: PAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Tommaso Gori, Professor, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PAN-1
Record Dates: First submitted 2012-10-18; First posted 2012-10-24 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Endothelial Function
Keywords: endothelial function; sympathetic nervous system

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Myogenic activation (Active Comparator): Subjects will undergo endothelial function assessment at rest and, after a 45 minutes pause, 1 minute after begin of myogenic activation
  Interventions: Procedure: Myogenic activation
- Cold pressure test (Active Comparator): Subjects will undergo endothelial function assessment at rest and, after a 45 minutes pause, 1 minute after begin of cold pressure test
  Interventions: Procedure: Cold pressure test
- mental stress (Active Comparator): Subjects will undergo endothelial function assessment at rest and, after a 45 minutes pause, 1 minute after begin of mental stress
  Interventions: Procedure: Mental stress
- Control (Active Comparator): Control visit - no intervention performed - subjects will undergo endothelial function measurement twice at a distance of 45 minutes
  Interventions: Other: no intervention

INTERVENTIONS:
Procedure: Mental stress — Subjects will be asked to perform complex mathematic operations at a very fast pace
  Arms: mental stress
Other: no intervention — control visit
  Arms: Control
Procedure: Myogenic activation — A pneumatic cuff will be inflated to suprasystolic pressure around both thighs and the subjects will be asked to perform plantar flexion exercises.
  Arms: Myogenic activation
Procedure: Cold pressure test — A hand will be placed in ice-cold water.
  Arms: Cold pressure test

SUMMARY:
The purpose of this study is to determine whether interventions aimed at increasing sympathetic tone modify endothelial function measures as assessed by the measurement of flow-mediated dilation (FMD) and constriction (FMC). The investigators hypothesize that the three interventions under study will increase FMC while causing a blunting in FMD.

Further, the investigators plan to study the circadian variability of FMC and FMD. The investigators hypothesize a peak of FMD in the late hours of the day and a peak of FMC in the early hours.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers with no cardiovascular risk factor, no current disease, normal laboratory parameters and ECG.

Exclusion Criteria:

* any active disease

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in FMD in response to sympathetic activation | Change in FMD before versus 1 Minute after begin of intervention
  Flow-mediated dilation will be measured at rest and during each of the interventions.

SECONDARY OUTCOMES:
Change in FMC during sympathetic activation | Change in FMC before versus 1 minute after begin of each intervention
  Change in Flow-mediated constriction induced by each of the interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Gori, MD PhD, Principal Investigator — University Medical Center Mainz
Locations (1):
- University Medical Center Mainz, Mainz, Rhineland-Palatinate, Germany